CLINICAL TRIAL: NCT00444262
Title: Study Multicentric, Randomised, in Duplicate Blind Person of the Impact of a Per Operatory Strategy of Optimization of the Cardiac Output on the Forecast of the Old Subjects Operated for Fracture of the Upper End of the Femur " FRACTALE "
Brief Title: Stroke Volume Optimisation in Patients With Hip Fracture
Acronym: FRACTALE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: termination of the study due to difficulties to include patients
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fresenius Kabi (Industry); GAMIDA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P051009-AOM 05086
Record Dates: First submitted 2007-03-06; First posted 2007-03-07 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-06

CONDITIONS: Hip Fractures
Keywords: Hemodynamic optimisation; Esophageal Doppler; Hydroxy ethyl starch; Hip fracture; Outcome; Elderly subjects (≥ 70 year old); General anesthesia
MeSH Terms: conditions — Hip Fractures | interventions — HES 130-0.4

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): conventional treatment
  Interventions: Drug: VOLUVEN and others solute
- 2 (Experimental): stroke volume optimisation
  Interventions: Procedure: hemodynamic optimisation guided using esophageal Doppler

INTERVENTIONS:
Procedure: hemodynamic optimisation guided using esophageal Doppler — hemodynamic optimisation guided using esophageal Doppler
  Arms: 2
Drug: VOLUVEN and others solute — VOLUVEN and others solute
  Arms: 1

SUMMARY:
The aim of this study is to assess whether intra-operative fluid supplementation (to improve tissue perfusion) can reduce the incidence of postoperative complications in elderly patients with hip fracture.

DETAILED DESCRIPTION:
Rationale : Hip fracture patients frequently develop postoperative complications that increase their hospital length of stay and the cost of care. These complications are also associated with increased mortality. Perioperative tissue hypoperfusion may participate in the development of postoperative complications. Hypovolemia is secondary to many factors in hip fracture patients (including blood loss, fasting and dehydration) and can result in low cardiac output and tissue hypoperfusion. Two single-center, randomized, double-blind studies have demonstrated that peroperative fluid titration guided by esophageal Doppler measurements of stroke volume could improve patient outcome. Interpretation of these results was that such a stroke volume "optimisation" strategy could help the anesthesiologist give more fluids to his patient and reduce the risk of hypoperfusion without the risk of congestion, thereby reducing postoperative complications and improving patient outcome. We want to test the same hypothesis in a multicenter trial to confirm with a high level of proof the usefulness of this strategy. If previous results are confirmed, this could lead to a change in current anesthetic management of hip fracture patients and potentially have a very important economical impact on health costs.Goals : Primary endpoint is to demonstrate that colloid (Voluven®) titration, guided using esophageal Doppler estimation of stroke volume, during the surgical repair of hip fracture reduces the incidence of postoperative complications (composite criteria). Secondary endpoints in the "optimised group" include : 1) reduced delay to walk without help ; 2) increased number of days " out-of-hospital " at 3 months after the fracture ; and 3) reduced 1-year mortality.

ELIGIBILITY:
Inclusion criteria:

* Elderly subjects (≥ 70 year old) with hip fracture

Exclusion criteria:

* Patient or legal representative unwilling to give informed consent
* Patient with other trauma lesions associated to hip fracture
* Patient with esophageal disease or chronic dissection of the descending aorta (contra-indications to esophageal Doppler monitoring)
* Patient with known active neoplasia or with obvious metastatic hip fracture
* Allergy to hydroxy-ethyl starches
* Congenital hemostatic disorder

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 215 (Actual)
Dates: Start 2007-04; Primary Completion 2010-11 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
We expect a 30% reduction in the number of per- and post-operative complications observed during hospitalisation in acute care beds in the "optimised" subgroup with respect to "conventional" subgroup. Complications include: death, per-operative | during hospitalisation in acute care

SECONDARY OUTCOMES:
We will check if patients in the "optimised" group have:1) a reduction in the delay to walk without help2) more days " out-of-hospital " at 3 months 3) a reduction in 1-year mortality rate | at 3 months and at one year

CONTACTS AND LOCATIONS:
Overall Officials: bernard CHOLLEY, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (19):
- France (19):
  - Centre Hospitalier Universitaire de La Cote de Nacre, Caen, Calvados
  - Hopital Purpan, Toulouse, Haute Garonne
  - Hopital Antoine Beclere, Clamart, Hauts de Seine
  - Hopital D'Instruction Des Armees Percy, Clamart, Hauts de Seine
  - Hopital Beaujon, Clichy, Hauts de Seine
  - Hopital Lapeyronie, Montpellier, Herault
  - Hopital Lariboisiere, Paris, Paris
  - Hopital Saint Antoine, Paris, Paris
  - Hopital La Pitie Salpetriere, Paris, Paris
  - Fondation Saint Joseph, Paris, Paris
  - Hopital Cochin, Paris, Paris
  - Hopital Europeen Georges Pompidou, Paris, Paris
  - Hopital Bichat, Paris, Paris
  - Centre Hospitalier de Meaux, Meaux, Seine Et Marne
  - Centre Hospitalier Universitaire Rouen, Rouen, Seine Maritime
  - Hopital Avicenne, Bobigny, Seine Saint Denis
  - Hopital Henri Mondor, Créteil, Val de Marne
  - Hopital Bicetre, Le Kremlin-Bicêtre, Val de Marne
  - Centre Hospitalier Universitaire de Poitiers, Poitiers, Vienne